CLINICAL TRIAL: NCT00319007
Title: Adenoma-Carcinoma Sequence in the Ileal Pouch Anal Anastomosis in Patients With Familial Adenomatous Polyposis: Studies on Luminal and Mucosal Risk Factors and Chemoprevention
Brief Title: Influence of Sulindac and Probiotics on the Development of Pouch Adenomas in Patients With Familial Adenomatous Polyposis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 23266; KUN 2003-2911
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-08

CONDITIONS: Adenomatous Polyposis Coli
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Sulindac; Pharmaceutical Preparations; Probiotics; Inulin

INTERVENTIONS:
Drug: Sulindac (drug)
Drug: VSL#3 (probiotic)
Drug: Inulin (probiotic)

SUMMARY:
The purpose of this study is to determine whether sulindac and VSL#3 - inulin, either combined or alone, are effective in treating or preventing adenoma development in the ileal anal pouch in patients with familial adenomatous polyposis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically or genetically proven familial adenomatous polyposis
* Restorative proctocolectomy with ileal pouch anal anastomosis

Exclusion Criteria:

* Chronic or acute renal or hepatic disease
* History of oesophageal, gastric or duodenal ulcers
* Known hypersensitivity to sulindac
* Daily use during the last three months of:
* Aspirin
* Non-Steroidal Anti-Inflammatory Agents
* Probiotics

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Study Completion 2006-12

PRIMARY OUTCOMES:
Pouch mucosal proliferation index at 0, 1 and 2 months
Pouch mucosal apoptosis index at 0, 1 and 2 months

SECONDARY OUTCOMES:
Pouch mucosal Glutathione S transferases activity and isoenzyme levels at 0, 1 and 2 months
Faecal genotoxicity at 0, 1 and 2 months
Faecal cytotoxicity at 0, 1 and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Fokko M Nagengast, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands